CLINICAL TRIAL: NCT00105625
Title: Immunocompetency and Nutritive Status in Inpatient Gero-Rehabilitation
Brief Title: VA Nutrition Study on Immune Function
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: University of Oklahoma (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: NRI 99-340; OUHSC GCRC 0024
Record Dates: First submitted 2005-03-16; First posted 2005-03-17 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2008-06

CONDITIONS: Malnutrition; Infection; Nosocomial Infection
Keywords: Geriatrics; Nutrition; Immune function; Infection; Rehabilitation; Inpatient
MeSH Terms: conditions — Malnutrition; Infections; Cross Infection

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1

SUMMARY:
Hospital-acquired infections can occur five times as frequently in rehabilitation patients than in other hospital admissions. We postulate that this high infection rate may be due to nutritional problems frequently experienced in these patients. In this study, we examine the role of nutrition in inpatient geriatric rehabilitation patients' immune function and infection rates.

DETAILED DESCRIPTION:
Background:

Hospital-acquired infections can occur five times as frequently in rehabilitation patients than in other hospital admissions. We postulated that this high infection rate may be due to nutritional problems frequently experienced in these patients. In this study, we examined the role of nutrition in inpatient geriatric rehabilitation patients' immune function and infection rates.

Objectives:

We examined immunologic correlates of nutritional status in elderly veterans hospitalized for extended periods of inpatient rehabilitation. We tested the hypotheses that geriatric rehabilitation inpatients who receive standard clinical and dietary care: 1) experience deficiencies in nutrients important to immune function while they are hospitalized; and 2) those patients deficient in nutrients important for immune function experience higher infection rates.

Secondary objectives included: 1) identifying nutritional and physiological factors that might lead to immune function deficiencies and infection; and 2) developing a clinical assessment model of malnutrition that can be used to assess immune function in geriatric rehabilitation inpatients.

Methods:

In this descriptive cohort study, to test Hypothesis 1, we collected data to describe, over time, in 100 non-acute elderly patients receiving longer-term inpatient rehabilitation care, trends in and relationships among: 1) caloric, protein, and immunologically-relevant micronutrient intake; 2) body composition, metabolism, and biochemical indices of nutritional status; 3) humoral and cell mediated immunity; and 4) infection. To test Hypothesis 2, we collected data to examine differences in infection rates in adequately versus inadequately nourished patients. Secondarily, our study was conducted to examine the relationship of patients' eating, their nutritional status, and their immune function over time.

Status:

Project data collection activities have been completed. A total sample size of 100 patients completed the study protocol. No study-related serious adverse events occurred during study implementation. As declared above, while data analysis activities have been initiated as planned, no study results or findings are ready to report at this time.

ELIGIBILITY:
Inclusion Criteria:

Patients must be in inpatient rehabilitation, be > 55 years old, and must not suffer any of the following: on active antibiotics; chart documented malignancy, immunodeficiency (HIV, steroid treatment, plasma cell dyscrasia), advanced CHF or malabsorption syndromes (inflammatory bowel diseases such as colitis or Crohn's disease, celiac sprue, gastrectomy, bowel resection, irritable bowel syndrome, complicated diverticulitis, internal fistulae) affecting nutritional status; anemia (Hct<25%), renal failure (serum creatinine > 3.0 mg/dl), liver failure (alk phosp >3x norm or bilirubin >10mg/100ml); estimated LOS <3 months; unable to comply with study procedures.

Exclusion Criteria:

known pre-existing infection requiring antibiotic treatment (e.g. TB, osteomyelitis, SBE) chart documented malignancy, immunodeficiency (e.g. HIV infection, steroid treatment, plasma cell dyscrasia), advanced CHF or malabsorption syndromes (inflammatory bowel diseases such as colitis or Crohn's disease, celiac sprue, gastrectomy, bowel (ileal) resection, irritable bowel syndrome, complicated diverticulitis, or internal fistulae) directly affecting nutritional status documented anemia (Hct <25%), renal (serum creatinine >3.0 mg/dl), or liver failure (SGPT or alkaline phosphatase >3 times normal or bilirubin >10mg/100mL).

estimated admission <3 months or noncompliance with study procedures (unable/unwilling to perform study procedures)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2003-03; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonelle E. Wright, PhD MSN BSN, Principal Investigator — Oklahoma City VA Medical Center, Oklahoma City, OK
Locations (1):
- Oklahoma City VA Medical Center, Oklahoma City, OK, Oklahoma City, Oklahoma, United States